CLINICAL TRIAL: NCT01023516
Title: A 12-Week, Randomised, Double-Blind, Placebo-Controlled, Parallel Group, Multinational, Phase IIb Study to Evaluate the Efficacy and Safety of 60mg AZD9668 Administered Orally Twice Daily to Subjects With Chronic Obstructive Pulmonary Disease (COPD) on Treatment With Budesonide/Formoterol
Brief Title: Efficacy and Safety of Twice Daily 60mg AZD9668 in COPD for 12 Weeks in Patients on Background Budesonide/Formoterol
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D0520C00020
Record Dates: First submitted 2009-12-01; First posted 2009-12-02 (Estimated); Results first posted 2012-08-03 (Estimated); Last update posted 2012-08-03 (Estimated); Status verified 2012-06

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Chronic; obstructive; pulmonary; lung; respiratory disease; efficacy; placebo-controlled; COPD; FEV1; St Georges Respiratory Questionnaire
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchiolitis Obliterans Syndrome; Respiration Disorders | interventions — N-((5-(methanesulfonyl)pyridin-2-yl)methyl)-6-methyl-5-(1-methyl-1H-pyrazol-5-yl)-2-oxo-1-(3-(trifluoromethyl)phenyl)-1,2-dihydropyridine-3-carboxamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: AZD9668
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD9668 — 2 x 30 mg oral tablets bd for 12 weeks
  Arms: 1
Drug: Placebo — 2 x matched placebo to oral tablet bd for 12 weeks
  Arms: 2

SUMMARY:
The primary objective is to evaluate the efficacy of AZD9668 compared with placebo in symptomatic COPD patients by assessing the effects on lung function and symptoms of COPD

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD with symptoms over 1 year
* FEV1/FVC < 70% and FEV1 >= 30 and < 80 % of predicted post-bronchodilator
* Symptomatic COPD for a total of 7 days in the two weeks prior to randomisation
* At least 1 COPD exacerbation from 4 weeks to 12 months before the screening visit

Exclusion Criteria:

* Past history or current evidence of clinically significant heart disease
* Current diagnosis of asthma
* Patients who require long term oxygen therapy
* Worsening of COPD requiring treatment with antibiotics, an increase in inhaled steroid dose and/or oral steroids within 4 weeks of study visit 1b

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 615 (Actual)
Dates: Start 2009-11; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Kuna, Professor, Principal Investigator — Samodzielny Publiczny ZOZ Uniwersytecki Szpital Kliniczny
Locations (66):
- Bulgaria (8):
  - Research Site, Lovech
  - Research Site, Pleven
  - Research Site, Plovdiv
  - Research Site, Rousse
  - Research Site, Sofia
  - Research Site, Stara Zagora
  - Research Site, Troyan Municipality
  - Research Site, Varna
- Czechia (9):
  - Research Site, Jihlava
  - Research Site, Jindřichův Hradec
  - Research Site, Kladno
  - Research Site, Krnov
  - Research Site, Nový Jičín
  - Research Site, Pardubice
  - Research Site, Prague
  - Research Site, Rokycany
  - Research Site, Třebíč
- Hungary (11):
  - Research Site, Balassagyarmat
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Deszk
  - Research Site, Győr
  - Research Site, Nyíregyháza
  - Research Site, Pécs
  - Research Site, Százhalombatta
  - Research Site, Szombathely
  - Research Site, Törökbálint
  - Research Site, Vásárosnamény
- Poland (16):
  - Research Site, Bialystok
  - Research Site, Gdynia
  - Research Site, Gorzow Wlkp
  - Research Site, Grodzisk Mazowiecki
  - Research Site, Jelenia Góra
  - Research Site, Katowice
  - Research Site, Kielce
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Piła
  - Research Site, Skierniewice
  - Research Site, Szczecin
  - Research Site, Tarnów
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Romania (5):
  - Research Site, Constanța, Constanța County
  - Research Site, Deva, Hunedoara County
  - Research Site, Bucharest, Romania
  - Research Site, Bucharest
  - Research Site, Iași
- Slovakia (17):
  - Research Site, Bardejov
  - Research Site, Bojnice
  - Research Site, Bratislava
  - Research Site, Dunajská Streda
  - Research Site, Humenné
  - Research Site, Košice
  - Research Site, Liptovský Hrádok
  - Research Site, Nové Mesto nad Váhom
  - Research Site, Nové Zámky
  - Research Site, Poprad
  - Research Site, Považská Bystrica
  - Research Site, Prešov
  - Research Site, Revúca
  - Research Site, Spišská Nová Ves
  - Research Site, Trnava
  - Research Site, Trstená
  - Research Site, Žilina

REFERENCES:
- [Derived] Leidy NK, Murray LT, Monz BU, Nelsen L, Goldman M, Jones PW, Dansie EJ, Sethi S. Measuring respiratory symptoms of COPD: performance of the EXACT- Respiratory Symptoms Tool (E-RS) in three clinical trials. Respir Res. 2014 Oct 7;15(1):124. doi: 10.1186/s12931-014-0124-z. PMID 25287629
- [Derived] Leidy NK, Murray LT, Jones P, Sethi S. Performance of the EXAcerbations of chronic pulmonary disease tool patient-reported outcome measure in three clinical trials of chronic obstructive pulmonary disease. Ann Am Thorac Soc. 2014 Mar;11(3):316-25. doi: 10.1513/AnnalsATS.201309-305OC. PMID 24432712
- [Derived] Kuna P, Jenkins M, O'Brien CD, Fahy WA. AZD9668, a neutrophil elastase inhibitor, plus ongoing budesonide/formoterol in patients with COPD. Respir Med. 2012 Apr;106(4):531-9. doi: 10.1016/j.rmed.2011.10.020. Epub 2011 Dec 23. PMID 22197578

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient enrolled 24 November 2009. Last patient completed 18 August 2010. Study conducted at 79 centres in 6 countries (Bulgaria, Czech Republic, Hungary, Poland, Romania, Slovakia).
Pre-assignment Details: 3- or 4-week run-in period on budesonide/formoterol twice daily to stabilise patients on maintenance therapy before randomisation. Patients already on budesonide/formoterol required a 3-week run-in period and patients on ICS as monotherapy or in combination with any long-acting bronchodilator required a 4-week run-in period.
Groups:
- 60 mg AZD9668: AZD9668 2x30 mg oral tablets twice daily (bid) for 12 weeks
- Placebo: Matched Placebo Tablets
Period: Overall Study
Arm/Group | 60 mg AZD9668 | Placebo
Started | 313 | 302
Completed | 289 | 284
Not Completed | 24 | 18
Not completed — Voluntary discontinuation | 7 | 5
Not completed — Adverse Event | 9 | 6
Not completed — Safety reason | 0 | 3
Not completed — Study-specific criteria | 4 | 2
Not completed — Incorrect enrolment | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 60 mg AZD9668 | Placebo | Total
Number analyzed (Participants) | 313 | 302 | 615
Age Continuous [Median (Full Range); unit: Years] | 62 [42 to 80] | 61 [41 to 79] | 61.5 [41 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 81 | 161
  Male | 233 | 221 | 454

OUTCOME MEASURES:

1. Primary Outcome: Baseline Pre-bronchodilator FEV1 (L)
Description: Forced expiratory volume in 1 second (FEV1) as a measure of lung function, measured before bronchodilator (salbutamol) use in the clinic.
Time Frame: Day 1
Population: The efficacy analysis set for each outcome measure includes those patients who received at least one dose of investigational product and for whom a baseline and at least one post-randomisation measurement is available for that outcome measure. Patients were analysed by to randomised treatment in accordance with the intention to treat principle.
Measure: Mean (Standard Deviation); unit: L
Arm/Group | 60 mg AZD9668 | Placebo
Number analyzed (Participants) | 309 | 301
L | 1.49 (0.539) | 1.44 (0.519)

2. Primary Outcome: End-value Pre-bronchodilator FEV1 (L)
Description: End of treatment value - week 12 for completers, otherwise Last Observation Carried forward (LOCF)
Time Frame: up to week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | 60 mg AZD9668 | Placebo
Number analyzed (Participants) | 309 | 301
L | 1.45 (0.015) [lower limit 0.015] | 1.43 (0.015) [lower limit 0.015]

3. Secondary Outcome: Post-bronchodilator FEV1 (L) - Baseline
Description: Forced expiratory volume in 1 second (FEV1) as a measure of lung function, measured after bronchodilator (salbutamol) use in the clinic.
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L
Arm/Group | 60 mg AZD9668 | Placebo
Number analyzed (Participants) | 310 | 300
L | 1.59 (0.530) | 1.56 (0.518)

4. Secondary Outcome: Post-bronchodilator FEV1 (L) - End-value
Description: End of treatment value - week 12 for completers, otherwise Last Observation Carried forward (LOCF)
Time Frame: up to week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | 60 mg AZD9668 | Placebo
Number analyzed (Participants) | 310 | 300
L | 1.56 (0.014) [lower limit 0.014] | 1.54 (0.015) [lower limit 0.015]

5. Secondary Outcome: Pre-bronchodilator FVC (L) - Baseline
Description: Forced vital capacity (FVC) as a measure of lung function, measured before bronchodilator (salbutamol) use in the clinic.
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L
Arm/Group | 60 mg AZD9668 | Placebo
Number analyzed (Participants) | 309 | 301
L | 2.98 (0.781) | 2.94 (0.806)

6. Secondary Outcome: Pre-bronchodilator FVC (L) - End-value
Description: End of treatment value - week 12 for completers, otherwise Last Observation Carried forward (LOCF)
Time Frame: up to week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | 60 mg AZD9668 | Placebo
Number analyzed (Participants) | 309 | 301
L | 2.94 (0.022) [lower limit 0.022] | 2.93 (0.022) [lower limit 0.022]

7. Secondary Outcome: Post-bronchodilator FVC (L) - Baseline
Description: Forced vital capacity (FVC) as a measure of lung function, measured after bronchodilator (salbutamol) use in the clinic.
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L
Arm/Group | 60 mg AZD9668 | Placebo
Number analyzed (Participants) | 310 | 300
L | 3.16 (0.787) | 3.12 (0.822)

8. Secondary Outcome: Post-bronchodilator FVC (L) - End-value
Description: End of treatment value - week 12 for completers, otherwise Last Observation Carried forward (LOCF)
Time Frame: up to week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | 60 mg AZD9668 | Placebo
Number analyzed (Participants) | 310 | 300
L | 3.11 (0.021) [lower limit 0.021] | 3.11 (0.021) [lower limit 0.021]

9. Secondary Outcome: Baseline Pre-bronchodilator FEV6 (L)
Description: Forced expiratory volume in 6 seconds (FEV6) as a measure of lung function, measured before bronchodilator (salbutamol) use in the clinic.
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L
Arm/Group | 60 mg AZD9668 | Placebo
Number analyzed (Participants) | 309 | 301
L | 2.68 (0.729) | 2.61 (0.714)

10. Secondary Outcome: End-value Pre-bronchodilator FEV6 (L)
Description: End of treatment value - week 12 for completers, otherwise Last Observation Carried forward (LOCF)
Time Frame: up to week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | 60 mg AZD9668 | Placebo
Number analyzed (Participants) | 309 | 301
L | 2.61 (0.019) [lower limit 0.019] | 2.61 (0.019) [lower limit 0.019]

11. Secondary Outcome: Baseline Post-bronchodilator FEV6 (L)
Description: Forced expiratory volume in 6 seconds (FEV6) as a measure of lung function, measured post after bronchodilator (salbutamol) use in the clinic.
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L
Arm/Group | 60 mg AZD9668 | Placebo
Number analyzed (Participants) | 310 | 300
L | 2.85 (0.724) | 2.79 (0.716)

12. Secondary Outcome: End-value Post-bronchodilator FEV6 (L)
Description: End of treatment value - week 12 for completers, otherwise Last Observation Carried forward (LOCF)
Time Frame: up to week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | 60 mg AZD9668 | Placebo
Number analyzed (Participants) | 310 | 300
L | 2.77 (0.017) [lower limit 0.017] | 2.78 (0.018) [lower limit 0.018]

13. Secondary Outcome: Baseline Pre-bronchodilator FEF25-75% (L/Sec)
Description: Forced expiratory flow between 25% to 75% of vital capacity (FEF25-75%) as a measure of lung function, measured before bronchodilator (salbutamol) use in the clinic.
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/sec
Arm/Group | 60 mg AZD9668 | Placebo
Number analyzed (Participants) | 307 | 301
L/sec | 0.60 (0.380) | 0.55 (0.324)

14. Secondary Outcome: End-value Pre-bronchodilator FEF25-75% (L/Sec)
Description: End of treatment value - week 12 for completers, otherwise Last Observation Carried forward (LOCF)
Time Frame: up to week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: L/sec
Arm/Group | 60 mg AZD9668 | Placebo
Number analyzed (Participants) | 307 | 301
L/sec | 0.57 (0.016) [lower limit 0.016] | 0.56 (0.016) [lower limit 0.016]

15. Secondary Outcome: Baseline Post-bronchodilator FEF25-75% (L/Sec)
Description: Forced expiratory flow between 25% to 75% of vital capacity (FEF25-75%) as a measure of lung function, measured after bronchodilator (salbutamol) use in the clinic.
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/sec
Arm/Group | 60 mg AZD9668 | Placebo
Number analyzed (Participants) | 310 | 299
L/sec | 0.64 (0.367) | 0.60 (0.333)

16. Secondary Outcome: End-value Post-bronchodilator FEF25-75% (L/Sec)
Description: End of treatment value - week 12 for completers, otherwise Last Observation Carried forward (LOCF)
Time Frame: up to week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: L/sec
Arm/Group | 60 mg AZD9668 | Placebo
Number analyzed (Participants) | 310 | 299
L/sec | 0.62 (0.016) [lower limit 0.016] | 0.61 (0.016) [lower limit 0.016]

17. Secondary Outcome: Pre-bronchodilator IC (L) - Baseline
Description: Inspiratory capacity (IC) as a measure of lung function, measured before bronchodilator (salbutamol) use in the clinic.
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L
Arm/Group | 60 mg AZD9668 | Placebo
Number analyzed (Participants) | 310 | 301
L | 2.21 (0.661) | 2.17 (0.661)

18. Secondary Outcome: Pre-bronchodilator IC (L) - End-value
Description: End of treatment value - week 12 for completers, otherwise Last Observation Carried forward (LOCF)
Time Frame: up to week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | 60 mg AZD9668 | Placebo
Number analyzed (Participants) | 310 | 301
L | 2.13 (0.024) [lower limit 0.024] | 2.14 (0.025) [lower limit 0.025]

19. Secondary Outcome: Post-bronchodilator IC (L) - Baseline
Description: Inspiratory capacity (IC) as a measure of lung function, measured after bronchodilator (salbutamol) use in the clinic.
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L
Arm/Group | 60 mg AZD9668 | Placebo
Number analyzed (Participants) | 310 | 299
L | 2.33 (0.718) | 2.30 (0.665)

20. Secondary Outcome: Post-bronchodilator IC (L) - End-value
Description: End of treatment value - week 12 for completers, otherwise Last Observation Carried forward (LOCF)
Time Frame: up to week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | 60 mg AZD9668 | Placebo
Number analyzed (Participants) | 310 | 299
L | 2.30 (0.023) [lower limit 0.023] | 2.27 (0.023) [lower limit 0.023]

21. Secondary Outcome: PEF - Baseline Measured by Patient at Home (L/Min) in the Morning
Description: Peak Expiratory Flow (L/min) as a measure of lung function, measured at home by the patient each morning. Baseline is the mean of last 10 days of data before start of treatment.
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | 60 mg AZD9668 | Placebo
Number analyzed (Participants) | 312 | 301
L/min | 215.60 (98.406) | 213.24 (96.803)

22. Secondary Outcome: PEF - End-value Measured by Patient at Home (L/Min) in the Morning
Description: Peak expiratory flow (PEF)
Time Frame: Last 6 weeks on treatment
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: L/min
Arm/Group | 60 mg AZD9668 | Placebo
Number analyzed (Participants) | 312 | 301
L/min | 208.68 (2.153) [lower limit 2.153] | 211.93 (2.189) [lower limit 2.189]

23. Secondary Outcome: FEV1 - Baseline Measured by Patient at Home (L) in the Morning
Description: Forced Expiratory Volume in 1 second (L) as a measure of lung function, measured at home by the patient each morning. Baseline is the mean of last 10 days of data before start of treatment.
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L
Arm/Group | 60 mg AZD9668 | Placebo
Number analyzed (Participants) | 312 | 301
L | 1.40 (0.546) | 1.34 (0.516)

24. Secondary Outcome: FEV1 - End-value Measured by Patient at Home (L) in the Morning
Description: Forced Expiratory Volume in 1 second (L)
Time Frame: Last 6 weeks on treatment
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | 60 mg AZD9668 | Placebo
Number analyzed (Participants) | 312 | 301
L | 1.32 (0.012) [lower limit 0.012] | 1.32 (0.012) [lower limit 0.012]

25. Secondary Outcome: EXACT - Baseline Total Score
Description: EXAcerbations of Chronic pulmonary disease Tool, patient questionnaire as a measure of respiratory symptoms (reported as units on a 0 (best health status) to 100 (worst possible status) scale). Baseline is the mean of last 10 days of data before start of treatment.
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 60 mg AZD9668 | Placebo
Number analyzed (Participants) | 311 | 300
units on a scale | 45.47 (9.683) | 46.01 (8.900)

26. Secondary Outcome: EXACT - End-value Total Score
Description: EXAcerbations of Chronic pulmonary disease Tool, patient questionnaire as a measure of respiratory symptoms (reported as units on a 0 (best health status) to 100 (worst possible status) scale).
Time Frame: Last 6 weeks on treatment
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 60 mg AZD9668 | Placebo
Number analyzed (Participants) | 311 | 300
units on a scale | 42.78 (0.473) [lower limit 0.473] | 43.07 (0.480) [lower limit 0.480]

27. Secondary Outcome: BCSS - Baseline Total Score
Description: Breathlessness, Cough and Sputum Scale, patient reported questionnaire as a measure of respiratory symptoms (reported on a 0 (best health status) to 12 (worst possible status) scale). Baseline is the mean of last 10 days of data before start of treatment.
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 60 mg AZD9668 | Placebo
Number analyzed (Participants) | 312 | 301
units on a scale | 5.26 (1.787) | 5.44 (1.765)

28. Secondary Outcome: BCSS - End-value Total Score
Description: Breathlessness, Cough and Sputum Scale, patient reported questionnaire as a measure of respiratory symptoms (reported on a 0 (best health status) to 12 (worst possible status) scale).
Time Frame: Last 6 weeks on treatment
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 60 mg AZD9668 | Placebo
Number analyzed (Participants) | 312 | 301
units on a scale | 4.68 (0.085) [lower limit 0.085] | 4.68 (0.086) [lower limit 0.086]

29. Secondary Outcome: Sputum Colour - Baseline
Description: Sputum Colour as assessed by the Bronkotest scale, reported on a scale from 1 - clear (best health status) to 5 - dark green (worst possible health status).
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 60 mg AZD9668 | Placebo
Number analyzed (Participants) | 300 | 298
units on a scale | 1.87 (0.901) | 1.88 (0.807)

30. Secondary Outcome: Sputum Colour - End Value
Description: Sputum Colour as assessed by the Bronkotest scale, reported on a scale from 1 - clear (best health status) to 5 - dark green (worst possible health status). End of treatment week 12
Time Frame: End of treatment week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 60 mg AZD9668 | Placebo
Number analyzed (Participants) | 300 | 298
units on a scale | 1.63 (0.042) [lower limit 0.042] | 1.70 (0.042) [lower limit 0.042]

31. Secondary Outcome: Use of Reliever Medication
Description: Daily average of number of inhalations of reliever medication
Time Frame: Last 6 weeks on treatment
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: inhalations
Arm/Group | 60 mg AZD9668 | Placebo
Number analyzed (Participants) | 310 | 299
inhalations | 3.40 (0.124) [lower limit 0.124] | 3.37 (0.126) [lower limit 0.126]

32. Secondary Outcome: Incremental Shuttle Walk Test - Baseline
Description: Endurance time (s)
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | 60 mg AZD9668 | Placebo
Number analyzed (Participants) | 312 | 301
seconds | 351 (119.5) | 352 (108.3)

33. Secondary Outcome: Incremental Shuttle Walk Test - End Value
Time Frame: Week 12 - visit 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: seconds
Arm/Group | 60 mg AZD9668 | Placebo
Number analyzed (Participants) | 297 | 287
seconds | 363.6 (3.39) [lower limit 3.39] | 363.7 (3.44) [lower limit 3.44]

34. Secondary Outcome: Endurance Shuttle Walk Test - Baseline
Description: Endurance time (s)
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | 60 mg AZD9668 | Placebo
Number analyzed (Participants) | 312 | 301
seconds | 419 (269.4) | 449 (292.9)

35. Secondary Outcome: Endurance Shuttle Walk Test - End Value
Description: Assessed at vist 6 -( last on treatment clinic visit)
Time Frame: Week 12 - visit 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: seconds
Arm/Group | 60 mg AZD9668 | Placebo
Number analyzed (Participants) | 299 | 286
seconds | 449.6 (10.49) [lower limit 10.49] | 459.9 (10.68) [lower limit 10.68]

36. Secondary Outcome: St George's Respiratory Questionnaire (COPD) - Overall Score at Baseline
Description: St George's Respiratory Questionnaire for Chronic Obstructive Pulmonary Disease, as a measure of Quality of Life (reported on a scale from 0 (best health status) to 100(worst possible status)).
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | 60 mg AZD9668 | Placebo
Number analyzed (Participants) | 295 | 280
Scores on a scale | 54.52 (16.863) | 54.87 (17.575)

37. Secondary Outcome: St George's Respiratory Questionnaire (COPD) - End-value Overall Score
Description: St George's Respiratory Questionnaire for Chronic Obstructive Pulmonary Disease, as a measure of Quality of Life (reported on a scale from 0 (best health status) to 100(worst possible status)).Questionaire assessed on vist 6 -( last on treatment clinic visit)
Time Frame: Measured Day 1 and 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | 60 mg AZD9668 | Placebo
Number analyzed (Participants) | 295 | 280
Scores on a scale | 49.89 (0.777) [lower limit 0.777] | 50.66 (0.796) [lower limit 0.796]

38. Secondary Outcome: Exacerbations - Clinic Defined
Description: Number of patients having a clinic defined disease exacerbation.
Time Frame: Duration of the the treatment period - 12 weeks
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | 60 mg AZD9668 | Placebo
Number analyzed (Participants) | 312 | 301
Participants | 22 | 29

ADVERSE EVENTS:
Arm/Group | 60 mg AZD9668 | Placebo
Serious Adverse Events (participants affected / at risk) | 9/313 | 14/302
Other Adverse Events (participants affected / at risk) | 0/313 | 0/302
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 60 mg AZD9668 (N=313) | Placebo (N=302)
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 0 | 2
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 1
ANGINA PECTORIS (Cardiac disorders) | 0 | 1
BUNDLE BRANCH BLOCK RIGHT (Cardiac disorders) | 1 | 0
CARDIAC FAILURE (Cardiac disorders) | 0 | 1
PNEUMONIA (Infections and infestations) | 1 | 3
POST PROCEDURAL INFECTION (Infections and infestations) | 0 | 1
PYELONEPHRITIS ACUTE (Infections and infestations) | 1 | 0
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
LARYNGEAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
LUNG SQUAMOUS CELL CARCINOMA STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
SYNCOPE (Nervous system disorders) | 0 | 0
RENAL COLIC (Renal and urinary disorders) | 0 | 1
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 4 | 1
ACUTE PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No